CLINICAL TRIAL: NCT01523951
Title: A Comparison of Topical Local Anaesthesia and Cooling to Reduce the Burning Pain During Capsaicin 8% Patch Application
Brief Title: Topical Local Anaesthesia and Cooling During Capsaicin 8% Patch Application
Acronym: LACCA
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Collaborators: Astellas Pharma GmbH (Industry)
Responsible Party: Principal Investigator, E. Knolle, MD, Ao.Univ.-Prof. Dr. Erich Knolle, Medical University of Vienna
Other Study IDs: 367/180-03/04; 2011-002264-25 (EudraCT Number)
Record Dates: First submitted 2012-01-29; First posted 2012-02-01 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Pain
Keywords: topical local anaesthesia; cooling; capsaicin 8%; epidermal nerve fiber density; treatment pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Skin biopsy
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy volunteers

SUMMARY:
Aim of the study is to demonstrate superiority of a continuous cooling of the skin over topical EMLA or placebo in reducing the burning pain during the application of capsaicin 8% patch ("Qutenza").

Secondary it will be tested, if the 2 different pre-treatments have an effect on the application pain within the first 24 hours, and if different pre-treatments have an effect on the reduction of the epidermal nerve fiber density (ENFD) 1 week after Qutenza application.

DETAILED DESCRIPTION:
According to literature, one of the most common adverse events of capsaicin 8% patch is a burning pain and a reversible erythema at the application site. In general it is recommended to apply a topical anesthetic one hour before capsaicin 8% patch application, or to treat the pain with cooling, NSAIDs or even opioids. Nevertheless, there is still only limited data available on the effects and side-effects. In this study it shall be tested if cooling the skin down for about 5-10 Celsius, immediately before Qutenza is applied, and continuing the cooling during the whole application time, results in a reliable prevention of the burning pain compared to pretreatment with topical anesthesia applied one hour in advance. This would lead to the assumption that the application pain is predominantly caused by a decrease of the threshold for heat pain beyond skin temperature and can therefore be prevented by a lowering of the skin temperature.

By ascertaining pain 24 hours after capsaicin 8% patch application and epidermal nerve fiber density (ENFD) 1 week after capsaicin 8% patch application it shall be proved if the different pretreatment methods do not change the secondary effects of capsaicin application.

If results turn out to be positive, it would be a massive relief with regard to time management and rescue medication.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers 18 ore more years old

Exclusion Criteria:

* dermatologic or neurologic injuries on both thighs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy volunteers
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2012-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
burning pain during the application of capsaicin 8% patch | 60 minutes

SECONDARY OUTCOMES:
application pain within the first 24 hours after application of capsaicin 8% patch | 24 hours
epidermal nerve fiber density(ENFD) | 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Spec. Anesthesia and Pain Therapy, Vienna, Vienna, Austria